CLINICAL TRIAL: NCT03533998
Title: Biomarkers in Prostate Cancer Treated With Salvage Radical Prostatectomy Following Failure of Focal Ablative Therapies
Brief Title: Biomarkers in Prostate Cancer Treated With SRP Following Failure of FAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: URO-04-2018
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tumor tissue of radical prostatectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ability of genomic biomarkers to Measuring tumour aggressiveness, and facilitate the selection of therapies in patients who had salvage radical prostatectomy after focal therapy and predict the risk of biochemical recurrence BCR after focal therapy or RP.

DETAILED DESCRIPTION:
Between 2007 and 2017, 30 patients underwent salvage radical prostatectomy SRP for recurrent localized PCa at our institution (Institute Mutual Montsouris). Primary radiotherapy, brachytherapy and whole-gland treatments were excluded, as to evaluate the true spectrum of morphologic changes caused by the focal emerging ablative modalities. Thirteen SRP after focal ablative therapies FAT (cryotherapy or high intensity focused ultrasound- HIFU or vascular-targeted photodynamic therapy- VTP) were identified from our prospective collected database. Genitourinary pathologists were provided clinical information related to prior therapies and immunohistochemical (IHC) markers were used in the diagnosis of limited primary PC on needle biopsy when necessary. Prostatectomy specimens were processed and the number of tumor foci, size of the dominant focus and pathological stage were recorded. Residual disease was graded according to the Gleason grading system. Treatment-related histologic changes were examined.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer treated with salvage radical prostatectomy following failure of focal ablative therapies

Exclusion Criteria:

* Primary radiotherapy, brachytherapy and whole-gland treatments

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate
Study Population: Between 2007 and 2017, 30 patients underwent salvage radical prostatectomy SRP for recurrent localized PCa at our institution (Institute Mutualiste Montsouris).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-05-31 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
ability of genomic biomarkers to Measuring tumour aggressiveness | molecular analyses
  Fragment of Paraffin specimen after RP will be used for the analyses by Biomarkers; MYC, PTEN protein loss, chromosome 8 alterations
  .

CONTACTS AND LOCATIONS:
Overall Officials: Qusay Mandoorah, resident, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France